CLINICAL TRIAL: NCT01122173
Title: A Prospective, Single Arm Study of the Hansen System for Introducing and Positioning RF Ablation Catheters in Subjects With Paroxysmal Atrial Fibrillation
Brief Title: Use of the Hansen Medical System in Patients With Paroxysmal Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hansen Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMP010
Record Dates: First submitted 2010-05-10; First posted 2010-05-13 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Atrial Fibrillation; Robotic Control; Remote Control
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Robotic catheter manipulation, Ablation (Experimental): To evaluate the safety and effectiveness of the family of Artisan guide catheters when used to remotely introduce and position commercially available cardiac RF ablation catheters to treat subjects with paroxysmal atrial fibrillation.
  Interventions: Device: Ablation

INTERVENTIONS:
Device: Ablation — Atrial fibrillation ablation procedure
  Other Names: Sensei X Robotic Catheter System; Artisan Control Catheter; RF Ablation Catheters

SUMMARY:
The purpose of this study is to assess the safety and performance of the Hansen Medical Sensei Robotic System and Artisan Catheter when used to robotically manipulate RF ablation catheters for the treatment of paroxysmal atrial fibrillation (irregular heartbeats originating in the upper chambers of the heart).

DETAILED DESCRIPTION:
Subjects who satisfy the inclusion and exclusion criteria will be treated with an RF ablation catheter and Artisan guide catheters controlled by the Sensei X Robotic Catheter System.

Subject will be followed for a period of one year post ablation procedure.

Follow up visit time frames will be conducted at 7-day, 30-day, 90-day, 180-day and 365-day.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with paroxysmal atrial fibrillation who have had two or more spontaneously terminating episodes of atrial fibrillation, that last longer than 30 seconds and shorter than 7 days, in the nine months prior to enrollment. At least one episode must be documented with EKG, TTM, Holter monitor, or telemetry.
2. Failure of at least one Class I - IV anti-arrhythmic drug (AAD) for PAF as evidenced by recurrent symptomatic PAF, or intolerable side effects due to AADs. AADs are defined in Appendix B.
3. Signed informed consent.
4. Age 18 years or older
5. Able and willing to comply with all pre-, post-, and follow-up testing and requirements.

Exclusion Criteria:

1. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
2. Previous ablation for atrial fibrillation.
3. Atrial fibrillation episodes that last less than 7 days and are terminated by cardioversion.
4. Previous valvular cardiac surgery procedure.
5. Cardiac artery bypass graft procedure within the previous 180 days.
6. Previous septal defect repair.
7. Expecting cardiac transplantation or other cardiac surgery within the next 180 days.
8. Coronary PTCA/stenting within the previous 180 days.
9. Documented left atrial thrombus on ultrasound imaging (TEE).
10. Documented history of a thrombo-embolic event within the previous 365 days.
11. Diagnosed atrial myxoma.
12. Presence of an implanted ICD.
13. Presence of permanent pacing leads.
14. Significant restrictive, constrictive, or chronic obstructive pulmonary disease or any other disease or malfunction of the lungs or respiratory system with chronic symptoms.
15. Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment in this study.
16. Women who are pregnant.
17. Acute illness or active infection at time of index procedure documented by either pain, fever, drainage, positive culture and/or leukocytosis (WBC > 11,000 mm3) for which antibiotics have been or will be prescribed.
18. Creatinine > 2.5 mg/dl (or > 221 µmol/L).
19. Unstable angina.
20. Myocardial infarction within the previous 60 days.
21. Left ventricular ejection fraction less than 40%
22. History of blood clotting or bleeding abnormalities.
23. Contraindication to anticoagulation medications.
24. Contraindication to computed tomography or magnetic resonance imaging procedures.
25. Life expectancy less than 1 year.
26. Enrollment in another investigational study.
27. Uncontrolled heart failure (NYHA class III or IV heart failure).
28. Presence of an intramural thrombus, tumor, or other abnormality that precludes catheter introduction or positioning.
29. Presence of a condition that precludes vascular access.
30. Left atrial size ≥ 50mm.
31. INR greater than 3.0 within 24 hours of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-07; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gallinghouse, M.D., Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Andrea Natale, M.D., Principal Investigator — Texas Cardiac Arrhythmia Research Foundation; Brenda Cayme, RN., BSN, Study Director — Hansen Medical, Inc.
Locations (13):
- United States (9):
  - Banner Heart Hospital, Mesa, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Saint Barnabas Heart Center, Livingston, New Jersey
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Texas Health Arlington Memorial/Heart Place, Arlington, Texas
  - Texas Cardiac Arrhythmia Research Foundation (TCARF), Austin, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - Univeristy of Virginia, Charlottesville, Virginia
- IKEM, Dept of Cardiology, Prague, Czechia
- Gentofte University Hospital, Hellerup, Denmark
- Hospital Universitario Madrid Montepríncipe, Madrid, Spain
- John Radcliff Hospital, Oxford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic Catheter Manipulation, Ablation
Started | 150
Completed | 141
Not Completed | 9
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — Left study for other reasons | 3

BASELINE CHARACTERISTICS:
Arm/Group | Robotic Catheter Manipulation, Ablation
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 92
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 137
  More than one race | 0
  Unknown or Not Reported | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety-Incidence of Major Complications
Description: The primary safety endpoint was defined as the incidence of major complications, including all early onset (within 7 days of the ablation procedure) major complications, and the incidence of esophageal injury or pulmonary vein stenosis through 180 days.
Time Frame: within 7 days of the ablation procedure nd the incidence of esophageal injury or pulmonary vein stenosis through 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Catheter Manipulation, Ablation
Number analyzed (Participants) | 150
Participants
  Responders | 132
  Failures | 13
  Unknown | 5

2. Primary Outcome: Effectiveness-Freedom From Symptomatic Atrial Fibrillation (AF), Atrial Flutter, and Atrial Tachycardia Episodes
Description: The primary effectiveness endpoint is chronic success as demonstrated by the freedom from symptomatic atrial arrhythmia from days 91 to 365.
Time Frame: 91 - 365 days after the inital ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Catheter Manipulation, Ablation
Number analyzed (Participants) | 150
Participants
  Responders | 45
  Failures | 60
  Unknown | 45

3. Secondary Outcome: Acute Procedural Success
Description: Acute procedural success is defined as the successful ablation of at least three of four pulmonary veins as shown by pulmonary vein entrance block per vein during the initial ablation procedure. A subject is considered to be an acute procedural failure if acute procedural success cannot be obtained by using the Hansen system and, as a result, manual manipulation is needed to complete the ablation procedure with the ablation catheter.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Catheter Manipulation, Ablation
Number analyzed (Participants) | 150
Participants
  Responders | 142
  Failures | 8

4. Secondary Outcome: Chronic Safety-Incidence of Major Complications
Description: Chronic safety is defined as the incidence of Major Complications during the period from 8 - 365 days following the initial ablation procedure (excluding pulmonary vein stenosis and atrio-esophageal fistula from 8 - 180 days, which are included in the primary safety endpoint). The incidence of pulmonary vein stenosis and atrioesophageal fistula is included during the period from 181 - 365 days.
Time Frame: 8 - 365 days post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Catheter Manipulation, Ablation
Number analyzed (Participants) | 150
Participants
  Responders | 134
  Failures | 16

ADVERSE EVENTS:
Time Frame: Adverse event data were collected one year following the procedure.
Arm/Group | Robotic Catheter Manipulation, Ablation
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 28/150
Other Adverse Events (participants affected / at risk) | 34/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Catheter Manipulation, Ablation (N=150)
Arrhythmia (Cardiac disorders) | 18 (24)
Angina pectoris (Cardiac disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Heart block (Cardiac disorders) | 1 (1)
Perforation of the cardiac muscle (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pulmonary effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Bleeding (requiring treatment other than applying pressure & bandage) (Vascular disorders) | 2 (2)
Pseudoaneurysm (Vascular disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Benign prostatic hypertrophy (Reproductive system and breast disorders) | 1 (1)
Arrhytmia Prophylaxis (Cardiac disorders) | 1 (1)
Atrial fibrilation (Cardiac disorders) | 1 (1)
Cardiac ablation (Cardiac disorders) | 3 (3)
Fluid overload (Vascular disorders) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Pharyngeal haematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retroperitoneal haematoma (Vascular disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Catheter Manipulation, Ablation (N=150)
Arrhythmia (Cardiac disorders) | 27 (42)
Infection (Infections and infestations) | 11 (13)

LIMITATIONS AND CAVEATS:
Following the acquisition of Hansen, a decision was made to terminate the study. The PMA previously planned to be submitted year end 2016 will not be submitted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-12-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT01122173/Prot_000.pdf
  • Statistical Analysis Plan (2013-06-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT01122173/SAP_001.pdf